CLINICAL TRIAL: NCT02494180
Title: A Prospective, Non-inferiority Randomized Double-blinded Trial Comparing Fentanyl and Midazolam vs Diazepam and Pethidine for Pain Relief During Oocyte Retrieval
Brief Title: A Non-inferiority Trial on Pain Relief During Oocyte Retrieval
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Collaborators: The University of Hong Kong (Other); Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, lydia lai, Associate Consultant, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KW/FR-15-021(83-22)
Record Dates: First submitted 2015-06-17; First posted 2015-07-10 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Infertility
Keywords: fentanyl; midazolam; pethidine; diazepam
MeSH Terms: conditions — Infertility | interventions — Fentanyl; Meperidine; Diazepam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: intravenous fentanyl, midazolam (Placebo Comparator): group A will be given intravenous 0.1mg fentanyl and 5mg midazolam prior oocyte retrieval
  Interventions: Drug: fentanyl; Drug: Midazolam
- B: intravenous pethidine, diazepam (Placebo Comparator): group B will be given intravenous 25mg pethidine, 5mg diazepam prior oocyte retrieval
  Interventions: Drug: pethidine; Drug: Diazepam

INTERVENTIONS:
Drug: fentanyl — arm A receiving iv fentanyl
  Arms: A: intravenous fentanyl, midazolam
Drug: pethidine — arm B receiving iv pethidine
  Arms: B: intravenous pethidine, diazepam
Drug: Diazepam — arm B receiving iv diazepam
  Other Names: valium
  Arms: B: intravenous pethidine, diazepam
Drug: Midazolam — arm A receiving iv midazolam
  Other Names: dormicum
  Arms: A: intravenous fentanyl, midazolam

SUMMARY:
The objective of the trial is to compare fentanyl and midazolam vs diazepam and pethidine in terms of the pain levels and post-operative side effects of TUGOR

DETAILED DESCRIPTION:
In-vitro fertilization / embryo transfer (IVF / ET) is a well-established method to treat various causes of infertility. It involves multiple follicular development, retrieval of oocytes and embryo transfer after fertilization. Egg retrieval at the majority of IVF units is performed through the transvaginal route under ultrasound guidance (TUGOR) [1]. During TUGOR, the needle has to pass through the mucosa in the vaginal vault in order to puncture the follicles in the ovary. The procedures are generally short, lasting about 20-30 minutes but are still painful without anaesthesia or analgesia.

Intravenous sedation with or without local anaesthesia is the most widely used method. Conscious sedation is a safe and cost-effective method of providing analgesia and anesthesia for TUGOR. [2] It is easy to administer in cooperative and motivated patients. It has a relatively low risk for adverse effects on oocyte and embryo quality and pregnancy rates. [3] Paracervical block (PCB) in conjunction with conscious sedation during TUGOR was shown to significantly reduce the pain during TUGOR when compared to PCB alone [4].

A Cochrane review on various methods of sedation and analgesia for pain relief during TUGOR has shown no single method or delivery system appeared superior for pregnancy rates and pain relief. [5] Most of the methods seemed to work well and the effect was usually enhanced by addition of another method such as pain relief with paracervical block. [6]

The investigators' reproductive centre has recently aligned with the Assisted Reproduction Centre of the University of Hong Kong (HKU). The investigators are using 0.1mg fentanyl and 5mg midazolam intravenously for pain relief in TUGOR at Kwong Wah Hospital (KWH) whereas 5mg diazepam and 25mg pethidine intravenously are being used in HKU. The investigators would like to compare fentanyl and midazolam vs diazepam and pethidine in terms of pain levels and post-operative side effects of TUGOR in this prospective non-inferiority randomized double-blinded trial. The investigators postulate there are no differences in the pain levels between two groups but the postoperative side effects may be different.

ELIGIBILITY:
Inclusion Criteria:

* presence of both ovaries;
* body mass index less than 30
* written informed consent and
* Chinese

Exclusion Criteria:

* IVF cycle converted from ovulation induction or intrauterine insemination cycles;
* patient requests general anaesthesia for TUGOR;
* history of drug sensitivity to lignocaine/fentanyl/midazolam/diazepam/pethidine;
* less than 3 dominant follicles present;
* dominant follicles present in one ovary only and
* TUGOR performed on one side only.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shui Fan Lai, Principal Investigator — Kwong Wah Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Started | 85 | 85
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [35 to 38] | 37 [35 to 38] | 37 [35 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 85 | 170
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 85 | 85 | 170
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Pain Level During Oocyte Retrieval
Description: The pain level will be scored using visual analogue scale 0-10, 0 = no pain, 10 =most painful
Time Frame: will be assessed within 4 hours of oocyte retrieval
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
score on a scale
  vaginal pain | 0 [0 to 2.5] | 4 [1 to 7]
  abdominal pain | 2.5 [0 to 5] | 5 [2.5 to 7.5]

2. Primary Outcome: Pain Level After Oocyte Retrieval
Description: The pain level will be scored using visual analogue scale 0-10, 0 = no pain, 10 =most painful
Time Frame: will be assessed within 4 hours of oocyte retrieval
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
score on a scale
  vaginal pain | 0 [0 to 2] | 0 [0 to 2.5]
  abdominal pain | 2.3 [0 to 2.8] | 2 [0 to 3]

3. Secondary Outcome: Percentage of Participants With Side Effects by Type
Description: side effects will be scored by yes or no
Time Frame: will be assessed within 4 hours of oocyte retrieval
Measure: Number; unit: percentage of participants
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
percentage of participants
  nausea | 2.4 | 7.1
  vomiting | 0 | 1.2
  dizziness | 16.5 | 4.7
  drowsiness | 8.2 | 3.5
  shortness of breath | 0 | 1.2

4. Secondary Outcome: Patient's Satisfaction on Oocyte Retrieval
Description: satisfaction will be scored from 0-3 (0=excellent, 1=satisfactory, 2=fair, 3=unsatisfactory)
Time Frame: will be assessed within 4 hours of oocyte retrieval
Measure: Number; unit: percentage of participants
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
percentage of participants
  excellent | 47.7 | 15.3
  satisfactory | 38.8 | 55.3
  fair | 11.8 | 22.4
  unsatisfactory | 4.7 | 7.1

5. Secondary Outcome: Clinical Pregnancy Rate
Description: presence of intrauterine sac in ultrasound after a positive pregnancy test
Time Frame: will be assessed within ten weeks of oocyte retrieval
Measure: Number; unit: percentage of participants
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
percentage of participants | 14.1 | 23.5

6. Secondary Outcome: Ongoing Pregnancy Rate
Description: positive fetal heart pulsation seen in ultrasound at eight weeks of gestation
Time Frame: will be assessed within ten weeks of oocyte retrieval
Measure: Number; unit: percentage of participants
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
percentage of participants | 12.9 | 21.2

7. Secondary Outcome: Patient's Satisfaction on Pain Relief
Description: satisfaction on pain relief will be scored at 0-10 (10 being most satisfied)
Time Frame: within 4 hours after retrieval
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
score on a scale | 8 [7 to 10] | 7 [6 to 9]

8. Secondary Outcome: Sedation Level
Description: S = sleeping, easily aroused; 1 = awake and alert; 2 = occasionally drowsy, easy to arouse; 3 = frequently drowsy, arousable, drifts off to sleep during conversation; 4 = somnolent, minimal or no response to stimuli
Time Frame: immediately after retrieval
Measure: Count of Participants; unit: Participants
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
Number analyzed (Participants) | 85 | 85
Participants
  1 | 15 | 52
  2 | 14 | 17
  3 | 16 | 4
  4 | 21 | 5
  S | 18 | 7
  missing data | 1 | 0

ADVERSE EVENTS:
Time Frame: within 18 days of hCG which is also the urine pregnancy test date
Arm/Group | A: Intravenous Fentanyl, Midazolam | B: Intravenous Pethidine, Diazepam
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02494180/Prot_SAP_000.pdf